CLINICAL TRIAL: NCT01882881
Title: Effects of Polyphenolic-rich Dark Chocolate/Cocoa and Almonds on Cardiovascular Disease Risk Factors
Acronym: CAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Almond Board of California (Other); The Hershey Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PKE 107
Record Dates: First submitted 2013-04-12; First posted 2013-06-21 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Chocolate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy American Control Diet (Active Comparator)
  Interventions: Other: Healthy American Control Diet
- Dark Chocolate/Cocoa Diet (Experimental)
  Interventions: Other: Dark Chocolate/Cocoa Diet
- Almond Diet (Experimental)
  Interventions: Other: Almond Diet
- Dark Chocolate/Cocoa + Almond Diet (Experimental)
  Interventions: Other: Dark Chocolate/Cocoa + Almond Diet

INTERVENTIONS:
Other: Healthy American Control Diet — The Control Diet will be comprised of the same foods as the test diets except for the isocaloric substitution of almonds and/or dark chocolate and cocoa for sources of saturated fat; an approximate 250 kcal substitution. In an effort to keep all the diets consistent (except for the specific foods to be tested), the Control Diet will be slightly higher in fiber (20-25g) and lower in cholesterol (~250 mg) than the typical consumption practices (15g and 278 mg, respectively).
  Arms: Healthy American Control Diet
Other: Dark Chocolate/Cocoa Diet — The Dark Chocolate/Cocoa Diet will include a daily hot cocoa beverage containing 11g of natural cocoa powder and 6 pieces of Hershey's Bliss Dark Chocolate (43g of dark chocolate). This amount of dark chocolate and cocoa will allow for the isocaloric substitution with 1.5oz almonds. The total diet will provide ~33% of calories from fat. The SFA (~12%) in the Dark Chocolate/Cocoa Diet will match that of the Control Diet and be slightly higher than the Almond Diet, however the saturated fat will be comprised largely of stearic acid from the dark chocolate; cholesterol will be ≤200 mg/day. The fiber in the Dark Chocolate/Cocoa Diet will be higher than both the Control and Almond Diets due to the fiber content of the dark chocolate (~9g).
  Arms: Dark Chocolate/Cocoa Diet
Other: Almond Diet — The Almond Diet will include 1.5 oz of almonds daily and provide ~34% of calories from fat. The Almond Diet will be lower in SFA than the Control and Dark Chocolate/Cocoa Diets, containing ~ 8-9% calories from SFA. In addition, both almond containing diets will be slightly higher in MUFA and PUFA than the Control and Dark Chocolate/Cocoa Diets, as a result of the nutrient profile of the almonds. Cholesterol will be ≤200 mg/day; fiber will be increased compared to the Control Diet due to the inclusion of almonds.
  Arms: Almond Diet
Other: Dark Chocolate/Cocoa + Almond Diet — This diet is designed to test the additive effects of combining consumption of dark chocolate and cocoa with almonds. The diet will include the same hot cocoa beverage (11g) and dark chocolate pieces (43g) plus 1.5 oz of almonds. Additional high saturated fat foods are removed from the Control Diet to account for both the dark chocolate and almonds. As a result, the total fat will be similar to the other three test diets at ~34-35% and the SFA will match that of the Almond Diet at ~8-9%. The fiber content of this diet will be highest (~35g); cholesterol will remain ≤200 mg/day.
  Arms: Dark Chocolate/Cocoa + Almond Diet

SUMMARY:
The purpose of this study is to investigate the individual and combined effects of dark chocolate/cocoa and almonds on lipids, lipoproteins, antioxidant defense, lipid peroxidation, phenolic acids, inflammatory status, blood pressure and arterial health. It is hypothesized that dark chocolate/cocoa and/or almonds will favorably affect lipids, lipoproteins, antioxidants, inflammatory status, blood pressure and arterial health compared to a healthy American control diet; however, the effects will be greater when dark chocolate/cocoa and almonds are consumed together versus consumption of each food individually.

ELIGIBILITY:
Inclusion Criteria:

* Overweight and obese (BMI ≥25, ≤40 kg/m2)
* Moderately elevated LDL-C between the 25-95th percentile from NHANES:

105-194 mg/dL for males; 98-190 mg/dL for females.

Exclusion Criteria:

* Tobacco use
* Systolic blood pressure ≥159 mm Hg
* Diastolic blood pressure ≥ 99 mm Hg
* A history of myocardial infarction, stroke, diabetes mellitus, liver disease, kidney disease, and thyroid disease (unless controlled on meds)
* Blood pressure or cholesterol-lowering medication use
* Refusal to discontinue intake of putative cholesterol-lowering supplements (e.g. psyllium, fish oil, soy lecithin, niacin, fiber, flax, stanols/sterols)
* Vegetarianism or dietary practices that are inconsistent with the test diets
* Nut allergies
* Refusal to discontinue nutritional supplements, herbs, or vitamins
* History of inflammatory gastrointestinal disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Lipid/lipoprotein change (standard panel) | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
  Total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides
24-hour ambulatory blood pressure change | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
Flow-mediated dilation change | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
Lipoprotein class and subclass change | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
  The VAP© Test provides a direct measure of the following lipid and lipoprotein classes and subclasses: LDL, Lp(a), IDL, LDL1, LDL2, LDL3, LDL4, HDL, HDL2, HDL3, VLDL, VLDL1+2, VLDL3, TC, TG, Non-HDL, Remnant Lipoproteins, ApoB100, and ApoA1.

SECONDARY OUTCOMES:
Serum C-reactive protein change | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
Serum insulin change | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
Serum glucose change | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
Plasma flavonoid change | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
LDL oxidation potential change (plasma) | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
  The ex vivo resistance of LDL to Cu2+-mediated oxidation will be determined.
Urinary F2α-isoprostane change | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
Plasma tocopherol change | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)

OTHER OUTCOMES:
PON1 activity change (serum) | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)
Ex vivo cholesterol efflux change (serum) | 0 wk, 4 wk, 10 wk, 16 wk, and 22 wk (at baseline and after each of the 4 diet periods)

CONTACTS AND LOCATIONS:
Overall Officials: Penny M. Kris-Etherton, PhD, RD, Principal Investigator — Penn State University
Locations (1):
- Penn State Clinical Research Center, Noll Lab, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Lee Y, Berryman CE, West SG, Chen CO, Blumberg JB, Lapsley KG, Preston AG, Fleming JA, Kris-Etherton PM. Effects of Dark Chocolate and Almonds on Cardiovascular Risk Factors in Overweight and Obese Individuals: A Randomized Controlled-Feeding Trial. J Am Heart Assoc. 2017 Nov 29;6(12):e005162. doi: 10.1161/JAHA.116.005162. PMID 29187388